CLINICAL TRIAL: NCT02991508
Title: A Randomized Double-blind Placebo-controlled Phase 1 Study on the Safety, Tolerability and Pharmacokinetics/-Dynamics of Escalating Single Intravenous Doses of ADRECIZUMAB (HAM8101) in Healthy Male Subjects
Brief Title: Adrecizumab Phase 1 Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Adrenomed AG (Industry)
Responsible Party: Principal Investigator, Peter Pickkers, Prof. dr., Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Adrecizumab-phase1; 2015-005671-24 (EudraCT Number)
Record Dates: First submitted 2016-07-01; First posted 2016-12-13 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Healthy Volunteers
Keywords: Adrecizumab; Phase 1 clinical trial; Adrenomedullin; Healthy volunteers; Monoclonal recombinant antibody
MeSH Terms: interventions — enibarcimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Vehicle (20 mM His/HCl pH 6.0)
  Interventions: Drug: Placebo
- Adrecizumab 0.5 mg/kg (Active Comparator): To assess the safety, tolerability and pharmacokinetics/-dynamics of single escalating doses of ADRECIZUMAB (0.5 mg/kg, 2,0 mg/kg and 8,0 mg/kg administered as single infusion over 1 hour) in healthy male subjects.
  Interventions: Drug: Adrecizumab
- Adrecizumab 2.0 mg/kg (Active Comparator): To assess the safety, tolerability and pharmacokinetics/-dynamics of single escalating doses of ADRECIZUMAB (0.5 mg/kg, 2,0 mg/kg and 8,0 mg/kg administered as single infusion over 1 hour) in healthy male subjects.
  Interventions: Drug: Adrecizumab
- Adrecizumab 8.0 mg/kg (Active Comparator): To assess the safety, tolerability and pharmacokinetics/-dynamics of single escalating doses of ADRECIZUMAB (0.5 mg/kg, 2,0 mg/kg and 8,0 mg/kg administered as single infusion over 1 hour) in healthy male subjects.
  Interventions: Drug: Adrecizumab

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo
Drug: Adrecizumab
  Arms: Adrecizumab 0.5 mg/kg; Adrecizumab 2.0 mg/kg; Adrecizumab 8.0 mg/kg

SUMMARY:
This is the first clinical trial with ADRECIZUMAB. The purpose of this clinical trial to identify safety and tolerability of different doses of ADRECIZUMAB in healthy volunteers.

DETAILED DESCRIPTION:
Adrenomedullin (ADM) is a natural occurring 52 amino acid peptide which is mainly expressed in endothelial and smooth muscle cells. ADM plasma levels are increased in patients with sepsis and related with severity of disease. ADM is a key regulator of vasotonus and of endothelial integrity in sepsis.

ADRECIZUMAB is an antibody against the N-terminus of ADM which only partially inhibits the bioactivity of ADM. Several septic animal studies have shown that administration of ADRECIZUMAB leads to reduced catecholamine demand, improved renal function, improved fluid balance and improved survival.

The administration of ADRECIZUMAB to rodents and non-human primates (NHP) has been tolerated very well. Single dose and repeated administrations over 14 days to rats and NHP in the GLP toxicology and safety study have not shown any clinical side-effects or histopathological findings.

Based on these data the starting dose for human beings should be 0.5 mg/kg ADRECIZUMAB as single infusion over 1 hour and should be increased up to 8 mg/kg.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent to participate in this trial prior to any study-mandated procedure.
2. Male subjects aged 18 to 35 years inclusive.
3. Subjects have to agree to use a reliable way of contraception with their partners from study entry until 3 months after study drug administration.
4. BMI between 18 and 30 kg/m², with a lower limit of body weight of 50 kg and a upper limit of 100 kg.
5. Healthy as determined by medical history, physical examination, vital signs, 12 lead electrocardiogram, and clinical laboratory parameters.

Exclusion Criteria:

1. Unwillingness to abstain from any medication, recreational drugs, anti-oxidant or vitamin supplements during the course of the study and within 7 days prior to the treatment day.
2. Unwillingness to abstain from smoking or alcohol 1 day prior to the treatment day and during the first 24 hours of the study.
3. Surgery or trauma with significant blood loss or blood donation within 3 months prior to the treatment day.
4. History, signs or symptoms of cardiovascular disease, in particular:

   * History of frequent vasovagal collapse or of orthostatic hypotension
   * Resting pulse rate ≤45 or ≥100 beats / min
   * Hypertension (RR systolic >160 or RR diastolic >90)
   * Hypotension (RR systolic <100 or RR diastolic <50)
   * Conduction abnormalities on the ECG consisting of a 1st degree atrioventricular block or a complex bundle branch block
   * Any chronic cardiac arrhythmias, except PAC's, PVC's
5. Renal impairment: plasma creatinine >120 µmol/L
6. Liver function tests (alkaline phosphatase, AST, ALT and/or γ-GT) above 2x the upper limit of normal.
7. History of asthma
8. Atopic constitution
9. CRP above 2x the upper limit of normal or clinically significant acute illness, including infections, within 2 weeks before administration of the study drug.
10. Treatment with investigational drugs or participation in any other clinical trial within 30 days prior to study drug administration.
11. Known or suspected of not being able to comply with the trial protocol.
12. Known hypersensitivity to any excipients of the drug formulations used. Inability to personally provide written informed consent (e.g. for linguistic or mental reasons) and/or take part in the study.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-05-23 (Actual); Primary Completion 2016-09-22 (Actual); Study Completion 2016-09-22 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability expressed in total number of treatment related (serious) adverse events | 3 months follow-up period
  Adverse events include: Clinically significant variation in vital signs compared to baseline (blood pressure and heart rate), local infusion reaction at site of i.v. IMP infusion, clinically significant changes in ECG compared to baseline and clinically significant deflections in laboratory parameters compared to baseline.

SECONDARY OUTCOMES:
Area under the curve (AUC) of free Adrecizumab (pharmacokinetics) | T=0 hours, T=0.25 hours, T=0.5 hours, T=1 hours, T=1.5 hours, T=2 hours, T=3 hours, T=4 hours, T=8 hours, T=24 hours, T=7 days, T=14 days, T=28 days, T=60 days, T=90 days.
Peak plasma concentration (Cmax) of free Adrecizumab (pharmacokinetics) | T=0 hours, T=0.25 hours, T=0.5 hours, T=1 hours, T=1.5 hours, T=2 hours, T=3 hours, T=4 hours, T=8 hours, T=24 hours, T=7 days, T=14 days, T=28 days, T=60 days, T=90 days.
Terminal t1/2 of free Adrecizumab (pharmacokinetics) | T=0 hours, T=0.25 hours, T=0.5 hours, T=1 hours, T=1.5 hours, T=2 hours, T=3 hours, T=4 hours, T=8 hours, T=24 hours, T=7 days, T=14 days, T=28 days, T=60 days, T=90 days.
Clearance of free Adrecizumab (pharmacokinetics) | T=0 hours, T=0.25 hours, T=0.5 hours, T=1 hours, T=1.5 hours, T=2 hours, T=3 hours, T=4 hours, T=8 hours, T=24 hours, T=7 days, T=14 days, T=28 days, T=60 days, T=90 days.
Volume of distribution of free Adrecizumab (pharmacokinetics) | T=0 hours, T=0.25 hours, T=0.5 hours, T=1 hours, T=1.5 hours, T=2 hours, T=3 hours, T=4 hours, T=8 hours, T=24 hours, T=7 days, T=14 days, T=28 days, T=60 days, T=90 days.
Ex vivo cytokine production | T=0 hours, T=1 hours, T=8 hours, T=7 days, T=14 days, T=28 days, T=90 days.
  Whole blood will be stimulated with LPS after which cytokine production will be determined by ELISA.
Blood levels of norepinephrin, epinephrine, dopamine and renin | T=0 hours, T=0.25 hours, T=0.5 hours, T=1 hours, T=1.5 hours, T=2 hours, T=3 hours, T=4 hours, T=8 hours, T=24 hours.
Blood levels of endothelin and pro-enkephalin. | T=0, T=0.25, T=0.5, T=1, T=1,5, T=2, T=3, T=4, T=8, T=24 hours. T=7, T=14, T=28, T=60, T=90 days.
Plasma levels of adrenomedullin and MR-proadrenomedullin | T=0, T=0.25, T=0.5, T=1, T=1,5, T=2, T=3, T=4, T=8, T=24 hours. T=7, T=14, T=28, T=60, T=90 days.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Pickkers, MD, PhD, Principal Investigator — Radboudumc department of Intensive Care
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided